CLINICAL TRIAL: NCT04573374
Title: Comparing the Outcome of Pulpotomy Using Biodentine and Portland Cement in Mature Cases With Irreversible Pulpitis: Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Youssef, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2020-09-17
Record Dates: First submitted 2020-09-27; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Irreversible Pulpitis
Keywords: irreversible pulpitis; pulpotomy; Biodentine; Portland cement
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodentine (Active Comparator): Biodentine (BD; Septodont, St Maur-des-Fosses, France) is a calcium silicate capping material. Biodentine is mixed according to manufacturer's instructions and placed in a 2-3 mm layer above the pulp tissue using an amalgam carrier and gently packed using a condenser. Initial setting is achieved after 12 minutes.
  Interventions: Procedure: Pulpotomy
- Portland cement (Active Comparator): Preparation of Portland cement: Industrial Portland cement is mixed with Bisthmus oxide or Barium sulphate radio-opacifier in a 3:1 ratio. The mix is sieved through silk sieve then sterilized in hot air oven at 135 ֯C for 2 hours. Portland cement is mixed in a 3:1 powder: distilled water ratio and placed in the pulp chamber and condensed against a moist cotton pellet. A small cotton pellet moistened with saline is placed in the pulp chamber against PC for 5 seconds to ensure water uptake then removed
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Pulpotomy — Pulpotomy is the term for removal of the coronal pulp with the intent of maintaining the vitality of the remaining radicular pulp tissue.
  Other Names: Vital pulp therapy

SUMMARY:
The aim of the study is to compare the treatment outcome of pulpotomy using Biodentine or Portland cement regarding success rate and post-operative pain.

DETAILED DESCRIPTION:
* Patients will be screened for eligibility through obtaining medical and dental histories together with clinical [visual, palpation, percussion, cold sensitivity testing and probing] and radiographic evaluations for the teeth.
* After ensuring eligibilty, profound local anesthesia of the tooth will be achieved using 4% Articaine with 1: 100000 epinephrine (Septodont. Saint-Maur-des-Fosses. France).
* Caries will be removed using a round, high-speed bur with adequate water cooling.
* Cases will be randomly divided into two groups according to pulpotomy material either: Biodentine or Portland cement. Biodentine is mixed according to manufacturer's instructions and placed in a 2-3 mm layer above the pulp tissue using an amalgam carrier and gently packed using a condenser. Initial setting is achieved after 12 minutes. Preparation of Portland cement: Industrial Portland cement is mixed with Bisthmus oxide or Barium sulphate radio-opacifier in a 3:1 ratio. The mix is sieved through silk sieve then sterilized in hot air oven at 135 ֯C for 2 hours. Portland cement is mixed in a 3:1 powder: distilled water ratio and placed in the pulp chamber and condensed against a moist cotton pellet. A small cotton pellet moistened with saline is placed in the pulp chamber against PC for 5 seconds to ensure water uptake then removed.
* Appropriate interim restoration will be done and checked throughout follow up period. Patients will be referred for final restoration after endpoint of research. A post-operative periapical radiograph is taken after interim restoration placement.
* Patients will be contacted by telephone by the same operator to record pain intensity (at 6, 12, 24, 48 and after 7 days).
* Clinical and radiographic evaluation is scheduled at 3 months postoperatively, and the outcome will be determined according to clinical and radiographic criteria. Clinical criteria include: absence of tenderness to palpation or percussion and the tooth is functional, normal mobility and probing pocket depth. Soft tissues around the tooth are normal with no swelling or sinus tract. Radiographic criteria include: absence of periapical pathosis evident on the radiograph such as root resorption, root canal calcification, furcal pathosis or new periapical rarefaction. In case of failure, the tooth will be treated endodontically and referred for final restoration.

ELIGIBILITY:
Inclusion Criteria:

* Exposed permanent teeth with mature roots.
* Asymptomatic irreversible pulpitis (no or mild symptoms) and Symptomatic irreversible pulpitis {spontaneous pain or pain exacerbated by cold stimuli and lasting for a few seconds to several hours (interpreted as lingering pain)} compared to contralateral normal teeth, and which could be reproduced using cold testing.
* Pre-operative pain assessed as none (but clinically exposed), moderate or severe on Numerical Rating Scale (NRS).
* The tooth is restorable and free from advanced periodontal disease.
* Soft tissues around the tooth are normal with no swelling or sinus tract.
* Vital bleeding pulp tissue should be present in all canals after pulpotomy.
* Age: more than 18 years

Exclusion Criteria:

* Immature teeth.
* Necrotic pulp and absence of bleeding upon exposure.
* Teeth unresponsive to cold stimulation, presence of sinus tracts or swelling, presence of periapical rarefaction, internal or external root resorption or root canal calcification on radiograph.
* Non-restorable teeth or teeth indicated for post and core restoration
* Teeth with severe periodontal disease.
* Any serious medical problem that prevented the patient from receiving treatment or attending follow-up visits. Pregnant or lactating female patients.
* Patients who used long-acting Non-steroidal anti-inflammatory drugs (NSAIDs) before treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Pulpotomy Success rate | 3 months
  Clinical and radiographic evaluation is scheduled at 3 months postoperatively, and the outcome will be determined according to clinical and radiographic criteria. Clinical criteria include: absence of tenderness to palpation or percussion and the tooth is functional, normal mobility and probing pocket depth. Soft tissues around the tooth are normal with no swelling or sinus tract. Radiographic criteria include: absence of periapical pathosis evident on the radiograph such as root resorption, root canal calcification, furcal pathosis or new periapical rarefaction. In case of failure, the tooth will be treated endodontically and referred for final restoration.
Pulpotomy success rate | 6 months
  Clinical and radiographic evaluation is scheduled at 6 months postoperatively, and the outcome will be determined according to clinical and radiographic criteria. Clinical criteria include: absence of tenderness to palpation or percussion and the tooth is functional, normal mobility and probing pocket depth. Soft tissues around the tooth are normal with no swelling or sinus tract. Radiographic criteria include: absence of periapical pathosis evident on the radiograph such as root resorption, root canal calcification, furcal pathosis or new periapical rarefaction. In case of failure, the tooth will be treated endodontically and referred for final restoration.
Pulpotomy success rate | 12 months
  Clinical and radiographic evaluation is scheduled at 12 months postoperatively, and the outcome will be determined according to clinical and radiographic criteria. Clinical criteria include: absence of tenderness to palpation or percussion and the tooth is functional, normal mobility and probing pocket depth. Soft tissues around the tooth are normal with no swelling or sinus tract. Radiographic criteria include: absence of periapical pathosis evident on the radiograph such as root resorption, root canal calcification, furcal pathosis or new periapical rarefaction. In case of failure, the tooth will be treated endodontically and referred for final restoration.

SECONDARY OUTCOMES:
Post-operative pain | 6, 12, 24, 48 hours and 1 week
  Patients will be contacted by telephone by the same operator to record pain intensity on Numerical Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Aya A Gamal, MSc, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awawdeh L, Al-Qudah A, Hamouri H, Chakra RJ. Outcomes of Vital Pulp Therapy Using Mineral Trioxide Aggregate or Biodentine: A Prospective Randomized Clinical Trial. J Endod. 2018 Nov;44(11):1603-1609. doi: 10.1016/j.joen.2018.08.004. Epub 2018 Oct 3. PMID 30292451
- [Background] Li Y, Sui B, Dahl C, Bergeron B, Shipman P, Niu L, Chen J, Tay FR. Pulpotomy for carious pulp exposures in permanent teeth: A systematic review and meta-analysis. J Dent. 2019 May;84:1-8. doi: 10.1016/j.jdent.2019.03.010. Epub 2019 Apr 11. PMID 30981748
- [Background] Danesh G, Dammaschke T, Gerth HU, Zandbiglari T, Schafer E. A comparative study of selected properties of ProRoot mineral trioxide aggregate and two Portland cements. Int Endod J. 2006 Mar;39(3):213-9. doi: 10.1111/j.1365-2591.2006.01076.x. PMID 16507075